CLINICAL TRIAL: NCT00017927
Title: A Study of the Effects of Pegvisomant on Growth Hormone Excess in McCune-Albright Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010197; 01-D-0197
Record Dates: First submitted 2001-06-20; First posted 2001-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-06

CONDITIONS: McCune Albright Syndrome; Polyostotic Fibrous Dysplasia
Keywords: Acromegaly; McCune-Albright Syndrome; IGF-1; Adenoma; Hyperplasia; MAS; Polyostotic Fibrous Dysplasia; PFD
MeSH Terms: conditions — Fibrous Dysplasia, Polyostotic; Acromegaly; Adenoma; Hyperplasia | interventions — pegvisomant

INTERVENTIONS:
Drug: Pegvisomant

SUMMARY:
This study will examine the effect of pegvisomant on growth hormone excess in patients with McCune-Albright syndrome (MAS). Patients with this disease have polyostotic fibrous dysplasia-a condition in which areas of normal bone are replaced with fibrous growth similar to scar tissue, abnormal skin pigmentation (birth marks) and precocious (early) puberty. About 10 percent of patients have excess growth hormone (GH). GH stimulates the production of another hormone called insulin-like growth factor 1 (IGF-1). Together, GH and IGF-1 affect bone growth. The excess of these hormones in MAS can cause overgrowth of the bones of the face, hands and feet, excess sweating, or increased height.

Pegvisomant is a synthetic drug that binds to cell receptors where GH would normally bind, thus preventing the naturally occurring hormone from stimulating IGF-1 and bone growth as it normally would. This study will see if pegvisomant will reduce blood levels of IGF-1 and mitigate the effects of growth hormone excess, including bone pain, bone turnover, hand and foot swelling and sweating, and abnormal levels of related hormones.

Patients who were screened for polyostotic fibrous dysplasia and MAS under NIH protocol 98-D-0145 and were found to have MAS with excess growth hormone are eligible for this 36-week study. The screening protocol includes a history and physical examination, blood and urine tests, hearing, eye and dental examinations, pain and physical function evaluations, endocrine and bone screening tests, various bone imaging studies, including magnetic resonance imaging (MRI) and computed tomography (CT) scans and bone biopsy in patients over 6 years old.

Participants in the current study will receive daily injections of either pegvisomant or placebo (an inactive substance) for 12 weeks, followed by a 6-week "washout" period with no drug. Then, patients who received placebo will be switched, or "crossed over," to receive pegvisomant for another 12 weeks, and those who received pegvisomant will receive placebo. This will be followed by another 6-week washout period. The drug and placebo will be injected under the skin, similar to insulin injections. Blood and urine tests will be done at the beginning of the study and repeated every 6 weeks until the study ends.

DETAILED DESCRIPTION:
McCune-Albright Syndrome (MAS) was originally described as the triad of polyostotic fibrous dysplasia of bone, cafe-au-lait skin pigmentation and precocious puberty. Other endocrine abnormalities have been identified in this disease. Growth hormone (GH) excess is associated with MAS and occurs in approximately 10% of the patients. Current therapies of MAS involve separate treatment for the bone and endocrine diseases. We propose to test the effectiveness of a novel GH receptor antagonist, pegvisomant at reducing the growth hormone excess in these patients. Secondarily we shall also assess the impact of pegvisomant therapy on the fibrous dysplastic bone lesions associated with the disease.

The subjects will be patients with MAS and non-suppressible growth hormone as determined by standard oral glucose tolerant testing (OGTT) and an elevated insulin-like growth factor-1 (IGF-I). It will be a randomized, blinded crossover design. The primary and secondary measures of efficacy will be: the normalization of serum (IGF-I), a reduction in signs and symptoms of growth hormone excess, and a net change in Insulin-like Growth Factor Binding Protein 3 (IGFBP-3). The effect of pegvisomant on the fibrous dysplastic bone activity in these patients will be determined by a net change in the levels of bone turnover markers.

ELIGIBILITY:
INCLUSION CRITERIA:

Diagnosis of PFD/MAS as required in Protocol 98-D-0145

Growth hormone excess will be determined as a non-suppressible serum growth hormone by oral glucose tolerance test (OGTT). The OGTT parameter will be serum GH greater than 2.0 ng/ml at 60 minutes after an oral load of 75g glucose.

Two consecutive and duplicate measurements of serum IGF-I level should be at least 1.3 times greater than the upper limit of normal (age and sex adjusted according to laboratory normal range).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2001-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chanson P, Dib A, Visot A, Derome PJ. McCune-Albright syndrome and acromegaly: clinical studies and responses to treatment in five cases. Eur J Endocrinol. 1994 Sep;131(3):229-34. doi: 10.1530/eje.0.1310229. PMID 7921205
- [Background] Shenker A, Weinstein LS, Moran A, Pescovitz OH, Charest NJ, Boney CM, Van Wyk JJ, Merino MJ, Feuillan PP, Spiegel AM. Severe endocrine and nonendocrine manifestations of the McCune-Albright syndrome associated with activating mutations of stimulatory G protein GS. J Pediatr. 1993 Oct;123(4):509-18. doi: 10.1016/s0022-3476(05)80943-6. PMID 8410501
- [Background] Mastorakos G, Mitsiades NS, Doufas AG, Koutras DA. Hyperthyroidism in McCune-Albright syndrome with a review of thyroid abnormalities sixty years after the first report. Thyroid. 1997 Jun;7(3):433-9. doi: 10.1089/thy.1997.7.433. PMID 9226216